CLINICAL TRIAL: NCT05931107
Title: Evaluation of the Effect of Stress Ball in Patients With Irritable Bowel Syndrome
Brief Title: Effect of Stress Ball on Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bedriye Cansu DEMİRKIRAN (Other)
Responsible Party: Sponsor-Investigator, Bedriye Cansu DEMİRKIRAN, PhD student, Ataturk University
Organization: Ataturk University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Cansutez
Record Dates: First submitted 2023-06-27; First posted 2023-07-05 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Irritable Bowel Syndrome; Quality of Life; Depression; Anxiety; Stress
Keywords: Irritable Bowel Syndrome; patient; stress ball; Depression; Anxiety; Stress; Quality of Life
MeSH Terms: conditions — Irritable Bowel Syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball practice group (Stress ball squeezing) (Experimental): Patient information form, IBS symptom severity score, IBS quality of life scale and Depression-Anxiety-Stress scale will be administered by the researcher using face-to-face interview technique (pre-test) to the patients in both groups.The patients in the experimental group will be told how to use the stress ball in the room in the outpatient clinic and each patient will be given a stress ball. The first sessions of the patients will be held together with the patient in the outpatient clinic. Patients will apply a stress ball (squeezing the stress ball) once a day at home. In order to ensure the continuity of the stress ball application, the phone numbers of the patients will be taken and a reminder message will be sent every day. The patients' IBS symptom severity score will be evaluated every week.The experimental group has to squeeze the stress ball for 10-15 minutes every day for 4 weeks.
  Interventions: Other: Stress ball practice group (Stress ball squeezing)
- Control group (No Intervention): Patients who come to the outpatient clinic will be met, information will be given about the research, and consent will be obtained from the patients who agree to participate in the research. The groups of the patients who meet the inclusion criteria will be determined according to the randomization list.
  Patient information form, IBS symptom severity score, IBS quality of life scale and Depression-Anxiety-Stress scale will be administered by the researcher using face-to-face interview technique (pre-test) to the patients in both groups.
  Stress ball attempts will not be made to the patients in the control group. Phone numbers of patients in this group will be taken. Patients' IBS symptom severity score will be evaluated every week.
  Patients in both groups will continue to use routine treatments for 4 weeks. After the research is completed, the patients in the control group will be given a stress ball according to their wishes and will be informed about its application.

INTERVENTIONS:
Other: Stress ball practice group (Stress ball squeezing) — The stress ball is made of round, colorful, high-quality silicone. A stress ball of medium hardness and 6 cm in diameter (suitable for adult use) will be used in the research. When it is loosened, it returns to its original state. In the experimental group, the patients are required to squeeze the ball once after counting to three, inhale each time they squeeze the ball, exhale when they loosen their grip, and focus only on the ball. The experimental group has to squeeze the stress ball for 10-15 minutes every day for 4 weeks.
  Arms: Stress ball practice group (Stress ball squeezing)

SUMMARY:
Objective: This study will be conducted to evaluate the effect of stress ball on symptom severity, quality of life, depression, anxiety and stress in patients with irritable bowel syndrome (IBS).

Material and Method: The data of the randomized controlled experimental study will be collected at the gastroenterology outpatient clinic of Erzurum City Hospital. A simple randomization list was created with the Random Allocation Software program and it will be carried out with a total of 56 patients diagnosed with IBS, including 28 experimental and 28 control groups. Patients in the experimental group were asked to squeeze the stress ball for at least 10 minutes every day for 4 weeks. No treatment will be applied to those in the control group. Patient information form, IBS symptom severity score, IBS quality of life scale, Depression-Anxiety-Stress scale will be used to collect research data.

Keywords: Irritable Bowel Syndrome, patient, stress ball, Depression, Anxiety, Stress, Quality of Life

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic biopsychosocial disorder characterized by recurrent abdominal pain, constipation and/or diarrhea, bloating, flatulence, and urgent defecation.The diagnosis of IBS is made using the Rome IV criteria. With the emergence of IBS symptoms, individuals' daily lives, work, sleep patterns, leisure time, eating habits, travels, sexual and social relationships are adversely affected. It is stated that anxiety and depression exacerbate IBS symptoms, impair quality of life, increase health service seeking behaviors, and increase health care use and costs.

This study will be conducted to evaluate the effect of stress ball on symptom severity, quality of life, depression, anxiety and stress in patients with irritable bowel syndrome (IBS).

Patients who come to the outpatient clinic will be met, information will be given about the research, and consent will be obtained from the patients who agree to participate in the research. The groups of the patients who meet the inclusion criteria will be determined according to the randomization list.

Patient information form, IBS symptom severity score, IBS quality of life scale and Depression-Anxiety-Stress scale will be administered by the researcher using face-to-face interview technique (pre-test) to the patients in both groups.

The patients in the experimental group will be given information on how to use the stress ball in the room in the outpatient clinic and a stress ball will be given to each patient. The first sessions of the patients will be held together with the patient in the outpatient clinic. Patients will apply a stress ball (squeezing the stress ball) once a day at home. The stress ball is made of round, colorful, high-quality silicone. A stress ball of medium hardness and 6 cm in diameter (suitable for adult use) will be used in the research. When it is loosened, it returns to its original state. In the experimental group, the patients are required to squeeze the ball once after counting to three, inhale each time they squeeze the ball, exhale when they loosen their grip, and focus only on the ball. In order to ensure the continuity of the stress ball application, the phone numbers of the patients will be taken and a reminder message will be sent every day. A 4-week record will be created and they will be asked to mark the data showing the amount of application each day to be allocated. The IBS symptom score will be evaluated by searching the prices of each week.

There will be no intervention in the control units. Phone numbers of patients in this group will be taken, and IBS symptom severity scores will be evaluated every week.

Patients in both groups will be called to the outpatient clinic at the end of the 4th week. IBS symptom severity score, IBS quality of life scale and Depression-Anxiety-Stress scale will be applied to the patients in the outpatient clinic (post test).

Patients in both groups will continue to use routine treatments for 4 weeks. After the research is completed, the patients in the control group will be given a stress ball according to their wishes and will be informed about its application.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with IBS according to Rome IV criteria,
* A score of 75 or higher (not in remission) on the IBS symptom severity score,
* Scoring 9 and below for depression (without depression), 7 and below for anxiety (without anxiety), and 14 and below for stress (without stress) on the Depression-Anxiety-Stress scale.
* are ≥18 years of age,
* Having no physical problems (any fracture, open wound and lack of muscle strength in the hand, wrist and arm) for squeezing the stress ball,
* No problem in communicating,
* IBS patients who accepted to participate in the study will be included in the study.

Exclusion Criteria:

* A score of 74 or less (in remission) on the IBS symptom severity score.
* A score of 9 and below for depression (without depression), 7 and below for anxiety (without anxiety), and 14 and below for stress (without stress) on the Depression-Anxiety-Stress scale.
* Having any physical disability (any fracture, open wound and lack of muscle strength in the hand, wrist and arm) to squeeze the stress ball,
* Patients who have problems communicating,
* Patients who wish to withdraw from the study will be excluded from the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-07-19 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome Symptom Severity Score, | Four weeks
  The IBS symptom severity score was developed to assess the severity of symptoms in IBS. The scale is widely used to monitor the progression and treatment of the disease. The IBS-SSS assesses the severity and duration of abdominal pain (abdominal pain, painful days), abdominal bloating (bloating), satisfaction with bowel habits (bowel habit), and quality of life. The scale consists of a total of 5 questions, each ranging from 0 to 100 points. The total score of the scale ranges from 0 to 500, and high scores indicate an increase in disease severity. In the scale, 0-74 points are classified as remission, 75-174 as mild, 175-299 as moderate, 300 points and above as severe severe IBS.

SECONDARY OUTCOMES:
Irritable Bowel Syndrome Quality of Life Scale | Four weeks
  Patrick et al. It was created by IBS to evaluate the quality of life in patients with IBS. In this scale, which was prepared for patients with irritable bowel syndrome, there are 5 Likert-type response options (1: Never, 2: Some, 3: Moderate, 4: A lot, 5: A lot). The scale consists of 8 sub-dimensions and 34 items; Sub-dimensions; dysphoria, activity , body image , health concern, food avoidance, social reaction , sexual and social relationship. Scores from each sub-dimension are calculated in itself. The overall score of the scale is determined by the total scores obtained from 34 items. The raw scores obtained from the scale sub-dimension and its total range between 34-170. Higher scale scores indicate that individuals' quality of life increases. The validity and reliability study in our country was carried out by Özgürsoy Uran et al.
Depression-Anxiety-Stress Scale | Four weeks
  The Turkish validity and reliability study of the scale developed by Lovibond and Lovibond was carried out by Bilgel and Bayram. The scale was a 4-point Likert scale type. The scale consists of 3 sub-dimensions (depression, anxiety, stress). Each sub-dimension consists of 14 items and there are 42 items in total. Depression items measure dissatisfaction, helplessness, worthlessness, loss of interest and low energy level. Anxiety items assess the individual's level of autonomic arousal, situational anxiety, subjective anxiety, and muscle response. Stress items are difficulty to relax, nervous stimulation, upset and boredom, discomfort, overreaction and intolerance. measures the level of symptoms. The total scores of the scale vary between 0 and 42 for each sub-dimension, and as the score increases, depression, anxiety and stress increase. In the scale, depression, anxiety and stress are divided into five categories as normal, mild, moderate, severe and very severe.

CONTACTS AND LOCATIONS:
Overall Officials: Ataturk University, Study Director — Ataturk University Faculty of Nursing / Erzurum
Locations (1):
- Erzurum City Hospital, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No